CLINICAL TRIAL: NCT04227392
Title: Effect of Vaginal Radiofrequency Therapy on Vaginal Laxity : Pilot Trial
Acronym: ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-1801-444-001
Record Dates: First submitted 2020-01-01; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Vaginal Laxity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): women who undergo radiofrequency therapy
  Interventions: Device: vaginal radiofrequency

INTERVENTIONS:
Device: vaginal radiofrequency — 2 sessions of vaginal radiofrequency therapy with 3 week interval. A session last 20 minutes.

SUMMARY:
To examine the efficacy and safety of radiofrequency therapy on vaginal laxity, The investigators enrolled 30 women with vaginal laxity. Radiofrequency therapy was consisted of 2 sessions with 3 week interval. A session included 20 minutes radiofrequency therapy on vaginal mucosa. Vaginal laxity score, female sexual function index (FSFI), female sexual distress scale (FSDS), vaginal pressure, adverse events were examined. Follow up period is 3 months.

ELIGIBILITY:
Inclusion Criteria:

* vaginal laxity score >= 3
* negative pregnancy test within 2 months

Exclusion Criteria:

* genital anomaly
* pelvic prolapse stage >= stage 3
* active genital infection
* vulvar pain or deformity
* disease related to sexual behavior
* current, chronic NSAIDs intake
* fever
* any acute illness
* cognitive disorder
* pacemaker insertion
* metal implants

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
change of vaginal laxity score from baseline | baseline - at 2nd therapy session (3week from baseline) - 1 month from 2nd therapy session - 3 month from 2nd therapy session
  subjective vaginal laxity

SECONDARY OUTCOMES:
change of FSFI score from baseline | baseline - 1 month from 2nd therapy session - 3 month from 2nd therapy session
  female sexual function index, higher is better
change of FSDS score from baseline | baseline - 1 month from 2nd therapy session - 3 month from 2nd therapy session
  female sexual distress scale, lower is better
change of vaginal pressure from baseline | baseline - at 2nd therapy session (3week from baseline) - 1 month from 2nd therapy session - 3 month from 2nd therapy session
  vaginal pressure measured with manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyenggi DO, South Korea